CLINICAL TRIAL: NCT06650774
Title: Comparison of the Effects of Nintedanib and Pirfenidone on Pulmonary Function Test Parameters and Radiological Findingsin Patients With Pulmonary Fibrosis
Brief Title: Comparison of the Efficacy of Pirfenidone and Nintedanipine in Pulmonary Fibrosis
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Olcay Ayçiçek, Asist Proof, Karadeniz Technical University
Other Study IDs: 2024/111
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
Keywords: Pulmonay Fibrosis; Pirfenidone; Nintedanib
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Group 1: Pirfenidone Group
- Group 2: Nintedanibe Group

SUMMARY:
The goal of this observational study is to compare the effects of pirfenidone and nintedanib on lung function and radiologic findings in fibrotic lung diseases. The main question it aims to answer is:

• Do these two drugs have equivalent effects on progression in patients with pulmonary fibrosis? If there is a comparison group: The investigators will compare patients with pulmonary fibrosis receiving pirfenidone with patients with pulmonary fibrosis receiving nintedanip.

The investigators will compare patients with pulmonary fibrosis receiving pirfenidone and patients with pulmonary fibrosis receiving nintedanip.

Pulmonary function test parameters at 3rd, 6th, 9th and 12th months and differences of 6 MWT parameters compared to baseline will be compared between the two groups.

DETAILED DESCRIPTION:
The data of patients who were started Pirfenidone or Nintedanib treatment with the diagnosis of Idiopathic Pulmonary Fibrosis or Progressive Pulmonary Fibrosis according to An Official ATS/ERS/JRS/ALAT Clinical Practice guideline and treated for at least one year in our department between January 1, 2010 and December 31, 2022 were retrospectively analyzed. The included patients had not previously used steroids or similar drugs for lung disease. The study was initiated after approval of the local ethics committee.

File information, pulmonary function test parameters and radiologic data, gender, age and comorbidity information of all patients were obtained from the hospital database. Pulmonary function tests were performed using a COSMED Quark 2021 model device. Patients were divided into two groups as nintedanib and pirfenidone group and both groups were compared in terms of progression in pulmonary function tests and radiologic findings within 1 year of diagnosis. For this purpose, the difference of pulmonary function test parameters (FVC (mL-%), FEV1 (mL-%), FEV1/FVC, FEF25-75 (mL-%), and 6-minute walk test values at the 3rd, 6th, 9th and 12th months of all patients from the baseline values at the time of diagnosis were analyzed and these differences were compared between the two groups.Thorax CT findings were also compared between the two groups for the presence of progression. Patients whose radiologic and PFT data at initial presentation were not available, patients whose treatment was discontinued before 1 year due to side effects or unresponsiveness or death, and patients who were switched between the two drugs before 1 year had elapsed were excluded from the study.

Statistical analysis Kolmogorov-Smirnov test was used to test the normal distribution of the continuous variables. The data characterized by a normal distribution are expressed as mean±standard deviation. Student's t-tests was used for the comparison of the data which had a normal distribution. Mann-Whitney-U test was used for the comparison of the non-normally distributed data. The discrete variables were compared using Chi-squared test. P <0.05 was considered to be statistically significant. The data were analyzed using the SPSS statistical software (version 13.01, serial number 9069728, SPSS Inc., Chicago).

ELIGIBILITY:
Inclusion Criteria:

* The patients who were started Pirfenidone or Nintedanib treatment with the diagnosis of Idiopathic Pulmonary Fibrosis or Progressive Pulmonary Fibrosis according to An Official ATS/ERS/JRS/ALAT Clinical Practice guideline and treated for at least one year in our department between January 1 2010 and December 31 2022 The included patients had not previously used steroids or similar drugs for lung disease.
* Patients aged 18 years who have not used steroids or similar medication after diagnosis

Exclusion Criteria:

* Patients whose radiologic and PFT data at initial presentation were not available -Patients whose treatment was discontinued before 1 year due to side effects or unresponsiveness or death
* Patients who were switched between the two drugs before 1 year had elapsed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who were started Pirfenidone or Nintedanib treatment with the diagnosis of Idiopathic Pulmonary Fibrosis or Progressive Pulmonary Fibrosis according to An Official ATS/ERS/JRS/ALAT Clinical Practice guideline and treated for at least one year in our department between January 1 2010 and December 31 2022 The included patients had not previously used steroids or similar drugs for lung disease
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Comparison of pulmonary function test parameters of pirfenidone and nintedanip groups after 1-year follow-up | January 1 2010 and December 31 2022
  SFT values at 3, 6, 9 and 12 months were compared with baseline values and the difference between the two groups was analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Olcay Aycicek, Asist Prof, Principal Investigator — 1. Karadeniz Technical University Faculty of Medicine, Department of Chest Diseases
Locations (1):
- 1. Karadeniz Technical University Faculty of Medicine, Department of Chest Diseases, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I prefer to leave it until after the publication of the article

REFERENCES:
- [Background] Johannson KA, Strambu I, Ravaglia C, Grutters JC, Valenzuela C, Mogulkoc N, Luppi F, Richeldi L, Wells AU, Vancheri C, Kreuter M; Erice ILD Working Group. Antacid therapy in idiopathic pulmonary fibrosis: more questions than answers? Lancet Respir Med. 2017 Jul;5(7):591-598. doi: 10.1016/S2213-2600(17)30219-9. PMID 28664861